CLINICAL TRIAL: NCT00084708
Title: A Phase I Study of Intravenous (IV) Calcitriol in Combination With ZD1839 (IRESSA®) in Refractory Solid Tumors
Brief Title: Calcitriol and Gefitinib With or Without Dexamethasone in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Marwan Fakih, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000365546; RPCI-RPC-0207
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Calcitriol; Dexamethasone; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: dexamethasone
Drug: gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Calcitriol may help tumor cells develop into normal cells. Dexamethasone may increase the effectiveness and decrease the side effects of gefitinib and calcitriol.

PURPOSE: This phase I trial is studying the side effects and best dose of calcitriol when given together with gefitinib or when given together with gefitinib and dexamethasone in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD), toxic effects, and tolerability of calcitriol alone and in combination with gefitinib with or without dexamethasone in patients with advanced solid tumors.

Secondary

* Determine the pharmacokinetics and pharmacodynamics of these regimens in these patients.
* Determine any tumor responses in patients treated with these regimens.

OUTLINE: This is a dose-escalation study of calcitriol.

* Stage 1: Patients receive calcitriol IV over 1 hour on days 1, 15, and 22 and oral gefitinib once daily on days 8-28 during course 1. For all subsequent courses, patients receive calcitriol IV over 1 hour on days 1, 8, 15, and 22 and oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of calcitriol with a fixed dose of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Stage 2: Patients receive calcitriol (beginning at 1 dose level below the MTD determined in stage 1) and gefitinib as in stage 1. Patients also receive oral dexamethasone once on the day before and twice on the day of each dose of calcitriol.

Cohorts 3-6 patients receive escalating doses of calcitriol with fixed doses of gefitinib and dexamethasone until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 21-36 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* No unstable or uncompensated hepatic disease

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min
* No prior hypercalcemia
* No kidney, ureteral, or bladder stones within the past 10 years
* No unstable or uncompensated renal disease

Cardiovascular

* Ejection fraction ≥ 30%
* No heart failure or significant heart disease
* No significant arrhythmias
* No myocardial infarction within the past 3 months
* No unstable angina pectoris
* No symptomatic congestive heart failure
* No other unstable or uncompensated cardiac disease

Pulmonary

* No evidence of clinically active interstitial lung disease

  * Chronic, stable, asymptomatic, radiographic changes allowed
* No other unstable or uncompensated respiratory disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study treatment
* Able to receive oral medication
* Willing to have serial skin biopsies
* No prior allergic reaction to compounds of similar chemical or biological composition to study drugs or other agents used in this study
* No ongoing or active infection
* No known severe hypersensitivity to gefitinib or any of its excipients
* No psychiatric illness or social situation that would preclude study compliance
* No other severe or uncontrolled systemic disease or concurrent illness that would preclude study participation
* No other significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* No other concurrent systemic glucocorticoid therapy

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Recovered from prior major surgery
* No prior nephrectomy

Other

* Recovered from all prior anticancer therapy
* More than 30 days since prior non-approved or investigational drugs
* More than 7 days since prior thiazides
* No concurrent administration of any of the following:

  * Combination antiretroviral therapy for HIV-positive patients
  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
  * Calcium supplements
  * Thiazides
  * Digoxin
* No other concurrent investigational or commercial anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-11; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States